CLINICAL TRIAL: NCT04466501
Title: A Comparative, Controlled Study to Evaluate the Performance of the ACR | LAB Urine Analysis Test System
Brief Title: ACR | LAB Urine Analysis Test System Evaluation of Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy.io Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-ACR | LAB-MC-02
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ACR LAB for Professional User (Experimental)
  Interventions: Device: ACR LAB

INTERVENTIONS:
Device: ACR LAB — The ACR | LAB is a prescription-only, nurse- or clinician-conducted in vitro diagnostic (IVD) device. The device combines a urine stick kit with an easy to use smartphone application using an image recognition algorithm.

SUMMARY:
The ACR LAB is a prescription-only, nurse- or clinician-conducted in vitro diagnostic (IVD) device. The test is for the qualitative and semi- quantitative detection of Albumin, Creatinine, and the Albumin-to- Creatinine Ratio. The device is composed of a kit and a smartphone application using an image recognition algorithm.

The degree of agreement of the ACR | LAB as compared to the comparator device will be tested. Urine samples will be tested by a separate professional user on each device.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-80 years of age;
* Subjects who are healthy or pregnant; or
* Subjects diagnosed with a disease that normally represents itself with an abnormal concentration of albumin:

  * Diabetes Type I/Type II,
  * Hypertension,
  * Any kidney disease,
  * Other relevant conditions.
* Subjects with any pathological findings which might be identified by the urine test (according to the physician discretion);
* Subject is capable and willing to provide informed consent;
* Subject has facility with both hands
* Subject is capable and willing to adhere to the study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance agreement of the ACR |LAB compared to the comparator device, tested by professional users. | 11 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Central Kentucky Research Associates, Lexington, Kentucky
  - AccuMed research associates, Garden City, New York